CLINICAL TRIAL: NCT04717622
Title: Investigation of Fever Suspected as a Zoonosis Using Advanced Diagnostic Technologies- a Prospective Cohort Study
Brief Title: Investigation of Fever Suspected as a Zoonosis Using Advanced Diagnostic Technologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Yael Yagel MD, Senior doctor, infectious diseases institute Soroka UMC, Soroka University Medical Center
Other Study IDs: SOR-20-0287-CTIL
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Brucellosis; Zoonotic Disease
MeSH Terms: conditions — Brucellosis; Zoonoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be kept without any processing or analysis of human DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Zoonosis including brucellosis and rickettsial infections are a major contributor to infectious morbidity in southern Israel. The Bedouins, a nomadic tribal population residing in the Negev area are notably exposed to domesticated animals including livestock, camels and companion animals, and their living conditions, especially with respect to poor sanitation in different Bedouin communities also expose them to rodents and disease vectors such as insects and arthropods. In this study, we aim to identify Bedouin patients arriving at the Soroka University Medical Center, a tertiary hospital un the Negev, with undifferentiated fever, suspected as a zoonosis.

We intend to use molecular methods to better diagnose the infectious agent using whole blood and serum samples, and when available other tissues or body fluid, and use next generation sequencing technology to deeply examine bacterial features such as virulence factors, and host pathogen interactions.

DETAILED DESCRIPTION:
This study aims to apply advanced technologies for the investigation of febrile illness in the Bedouin population, in order to improve laboratory diagnosis in terms of rapidity and sensitivity and to better our understanding of the pathophysiology of infectious diseases in the Bedouin population including various environmental exposures such as animal, water and waste and antibiotic exposure, as well as host-pathogen interactions associated with pathogen virulence, factors associated with chronicity and relapse, and response to treatment.

Study protocol:

Enrollment:

1. After screening, patients will be approached and offered the opportunity to participate in the study.
2. After signing of an informed consent patient will be interviewed and an enrollment questionnaire will be filled out.
3. If the patient is enrolled in the ED, blood, saliva, and stool samples will be collected. In case the patient presented with a rash or a skin lesion, a swab from an open lesion will be obtained.
4. If patient was enrolled after receiving antibiotics, we will also attempt to locate leftover blood samples that were drawn in the ED prior to receiving antibiotics.

Follow up:

* During hospitalization:

  * Seven days after hospitalization or on day of discharge (whichever comes first), an attempt will be made to obtain a second set of samples (blood, saliva, and stool), and clinical data will be drawn from the medical records regarding resolution of symptoms, antibiotic treatment, complications etc. In case of any surgical procedures done during the hospitalization period for diagnostic or therapeutic purposes (e.g. skin biopsy, bone biopsy, arthrocentesis, lumbar puncture), any leftover material deemed unnecessary for clinical purposes will be utilized for analysis.
  * During the hospitalization, the patients will be interviewed and a WASH (Water, Sanitation and Hygiene) questionnaire will be filled.
* Post-discharge ambulatory follow- up:

  * In the case of a scheduled follow up visit in the infectious disease clinic (or any other planned visit in the ambulatory service of SUMC), if blood sampling is performed, an attempt will be made to obtain whole blood and serum samples for research purposes. If study-designated blood sampling is not feasible, leftover material will be utilized for research purposes. If deemed clinically relevant, a follow up questionnaire will be filled out.
* Recurrent hospitalizations within the study period

  o In case of recurrent admission during the year after enrolment, the hospitalization will be assessed by the research team as "related" or "non-related" to the original diagnosis. If considered related to the studied disease or its complications, an attempt will be made to perform another blood sampling, and any leftover material from clinical sampling of other body sites (biopsies, surgical intervention or drainage) will be utilized for analysis. If deemed clinically relevant, a follow up questionnaire will be filled out. As recurrent hospitalization are analyzed as part of the study, they will not be considered serious adverse events (SAE).
* Six months after enrollment:

  o Telephone interview for establishing clinical outcomes (protocol attached in appendix).
* End of study period:

  * One year post enrollment, data regarding antibiotic use, recurrent hospitalizations, and long term complications will be collected from the patient's' medical files.

Sample collection:

Every patient enrolled in this study will undergo the following workup:

Blood sampling:

Whole blood and serum samples will be obtained at enrollment, and if possible, upon discharge and every planned ambulatory outpatient clinic visit or recurrent hospitalization. In case that the patient was enrolled during hospital stay due to a positive test result, any remaining leftovers from clinical non-research samples obtained prior to antibiotic treatment, will potentially be used for research purposes, as long as they are not needed for clinical use, and within the usual time frame of their storage in the relevant hospital lab. Maximum blood volume obtained for analysis at each time point will be 10 ml for adults, and 5 ml for children.

Other clinical sampling:

At enrolment, saliva and stool samples will be obtained for microbiological analysis including microbiome profiling, and any rash or wound sampling will also be analyzed by molecular and metagenomic methods for the diagnosis of the culprit pathogen.

Sample processing and analysis:

All samples will be stored at the Moran-Gilad lab, Faculty of Health Sciences, Ben-Gurion University of the Negev, for five years after enrolment. Processing of the samples will be done in batches, and not in real time therefore, will not produce any real-time data that could affect clinical decisions. The results of the analysis will not be available for the treating physician. For the purpose of bacterial genomic/metagenomic sequencing, DNA will be extracted from whole blood samples, and only microbial DNA will be identified and analyzed from the extracted material. No research on human DNA will be performed in this study. Bacterial isolates grown in standard cultures will be analyzed for further characterization (e.g. virulence). Brucella or other bacterial isolates identified through standard cultures will be further analyzed using in-vitro models including tissue culture for the analysis of host-pathogen interactions. Immune response in clinical samples will be analyzed for host inflammatory signals (e.g. gene expression, measurement of proteins). For the purpose of improving diagnostic capability, specific PCR testing for zoonoses (such as Brucella, Rickettsia, and Q fever, or others as needed) will be done on whole blood samples, attempting to examine their utility and concordance with other means of diagnosis, and compared to serological workup that will be performed using serum samples. All samples will be analyzed according to proper biosafety level and good laboratory practices.

Meta-data collection and patient information All patients will be asked to fill a questionnaire regarding the details of their current illness (attached in Hebrew and Arabic), and their living conditions and exposure to animals.

Metadata including demographic data, health status, including chronic medical illnesses, and prior hospitalizations, past history of zoonotic illnesses, will be collected from the medical records. During hospitalization the following parameters will be collected: vital signs including time till resolution of fever, lab testing and imaging results, and any surgical procedure or intensive care unit stay.

Data will also be collected from the patient's medical records during the year following enrollment to the study regarding factors associated with clinical outcomes including: recurrent hospitalizations, antibiotic consumption, follow up blood test results such as inflammatory markers, blood count, liver enzymes, and follow up serologic testing.

Study period and size This study aims to include a total of 500 patients, over three years, starting September 2020.

Ethical considerations and data security All patients enrolled in the study will be assigned a serial study number. All samples collected during this study will be labeled with the study number, and no other identifying information will be present on the collected samples. Files containing meta-data and questionnaires will also be labeled using study number. Informed consent forms containing identifying data will be kept in a locked office accessed only by the study team and a coding file matching identifying material with study numbers will be saved on a password-protected server on hospital computers. Identifying data will be used for the purpose of the follow-up phone interview at the end of the study period, and all information obtained will then be de-identified and stored using the study code. All data will be stored using REDCap secured web application.

ELIGIBILITY:
Inclusion Criteria:

* - Willing and able to provide informed consent (in case of children the legal guardian is willing to provide informed consent)
* All patients of Bedouin origin arriving at the SUMC ED during the study period with:
* fever >38.1 (either documented or reported), without an apparent infection source plus one of the following signs or symptoms
* Headache
* Rash
* Arthralgia, arthritis
* Weakness
* Myalgia
* epididymo-orchitis
* leukopenia, thrombocytopenia, elevated liver enzymes
* other findings suggestive of zoonotic infection
* Patients who were diagnosed with a zoonotic infection prior to or during hospital stay.

Exclusion Criteria:

* - Patients with an established source of infection other than zoonosis (such as urinary tract infection, pneumonia, upper respiratory tract infection), or a non-infectious cause of fever (malignancy, rheumatic disease etc.).
* Pregnant women
* Children weighing less than 6.5 kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of Bedouin origin presenting with undifferentiated fever to the emergency departments (ED) at Soroka University Medical Center (SUMC) (adults) or hospitalized (internal medicine or pediatrics) between September 2020 until October 2023 will be screened and those who meet the inclusion criteria will be offered the opportunity to enroll in this study
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-23 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of zoonotic infections | patients will be under follow up for 6 months after enrollment
  Molecular modes of diagnosis will be examined, in order to improve sensitivity and time to diagnosis
Clinical outcomes- relapse | patients will be under follow up for 6 months after enrollment
  Assessment of infection relapse within 6 months
Clinical outcomes- symptom resolution | patients will be under follow up for 6 months after enrollment, medical records will be reviewed for a year after enrollment
  time to resolution of symptoms
Clinical outcomes- antibiotic use | patients will be under follow up for 6 months after enrollment, medical records will be reviewed for a year after enrollment
  recurrent use of antibiotics during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Yael Yagel, MD, Study Director — Senior doctor, infectious diseases
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No